CLINICAL TRIAL: NCT04660812
Title: A Phase 1b/2, Open-Label, Randomized Platform Study Evaluating The Efficacy and Safety of AB928 Based Treatment Combinations in Patients With Metastatic Colorectal Cancer
Brief Title: An Open Label Study Evaluating the Efficacy and Safety of Etrumadenant (AB928) Based Treatment Combinations in Participants With Metastatic Colorectal Cancer.
Acronym: ARC-9
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arcus Biosciences, Inc. (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ARC-9; 2020-005386-13 (EudraCT Number)
Record Dates: First submitted 2020-12-03; First posted 2020-12-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — quemliclustat; zimberelimab; Bevacizumab; regorafenib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Etrumadenant + Zimberelimab + mFOLFOX-6 +/- Bevacizumab (Experimental): Participants will receive oral etrumadenant in combination with zimberelimab +mFOLFOX-6 +/-bevacizumab by IV infusion.
  Interventions: Drug: Etrumadenant; Drug: Zimberelimab; Drug: Bevacizumab; Drug: m-FOLFOX-6 regimen
- mFOLFOX-6 +/- Bevacizumab (Active Comparator): Participants will receive mFOLFOX-6 +/- bevacizumab by IV infusion.
  Interventions: Drug: Bevacizumab; Drug: m-FOLFOX-6 regimen
- Regorafenib (Active Comparator): Participants will receive oral regorafenib
  Interventions: Drug: Regorafenib
- AB680 + Etrumadenant + Zimberelimab (Experimental): Participants will receive oral etrumadenant in combination with AB680 + zimberelimab by IV infusion.
  Interventions: Drug: AB680; Drug: Etrumadenant; Drug: Zimberelimab

INTERVENTIONS:
Drug: AB680 — AB680 is a cluster of differentiated CD73 Inhibitor
  Arms: AB680 + Etrumadenant + Zimberelimab
Drug: Etrumadenant — Etrumadenant is a dual adenosine receptor (A2aR and A2bR) antagonist
  Other Names: AB928
  Arms: AB680 + Etrumadenant + Zimberelimab; Etrumadenant + Zimberelimab + mFOLFOX-6 +/- Bevacizumab
Drug: Zimberelimab — Zimberelimab is a fully human anti-PD-1 monoclonal antibody
  Other Names: AB122
  Arms: AB680 + Etrumadenant + Zimberelimab; Etrumadenant + Zimberelimab + mFOLFOX-6 +/- Bevacizumab
Drug: Bevacizumab — Bevacizumab is administered as part of standard chemotherapy regimen
  Arms: Etrumadenant + Zimberelimab + mFOLFOX-6 +/- Bevacizumab; mFOLFOX-6 +/- Bevacizumab
Drug: m-FOLFOX-6 regimen — mFOLFOX-6 regimen is administered as part of standard chemotherapy regimen
  Arms: Etrumadenant + Zimberelimab + mFOLFOX-6 +/- Bevacizumab; mFOLFOX-6 +/- Bevacizumab
Drug: Regorafenib — Regorafenib is administered as part of standard chemotherapy regimen
  Arms: Regorafenib

SUMMARY:
This randomized phase 1b/2 open-label study will evaluate the antitumour activity and safety of etrumadenant (AB928) treatment combinations in participants with metastatic colorectal cancer.

DETAILED DESCRIPTION:
This is a multicenter, open-label Phase 1b/2 study in participants with metastatic colorectal cancer that will assess the antitumour activity and safety of etrumadenant.

Approximately 250 participants will be enrolled to 1 of 3 cohorts:

Cohort A) etrumadenant + zimberelimab +mFOLFOX-6 +/-bevacizumab vs mFOLFOX-6 +/-bevacizumab

Cohort B) etrumadenant + zimberelimab +mFOLFOX-6 +/-bevacizumab vs regorafenib

Cohort C) chemotherapy-free combinations of etrumadenant + zimberelimab + other agents

The primary objective of this clinical study is to evaluate the safety of etrumadenant-based combination therapy in participants with metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants ≥ 18 years of age
* Histologically confirmed metastatic colorectal adenocarcinoma
* Must have at least 1 measurable lesion per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Life expectancy at least 3 months
* Adequate hematologic and end-organ function
* Negative HIV, Hep B and Hep C antibody testing
* Agreement to remain abstinent or use contraceptive measures with female partners of reproductive potential, and agreement to refrain from donating sperm, for 30 days after the last dose of etrumadenant, 90 days after the last dose of zim, 180 days after mFOLFOX-6 and 180 days after bev, whichever is longer.

  * Inclusion Criteria for Cohort A:
* Disease progression following not more than one prior line of treatment for mCRC that consisted of oxaliplatin or irinotecan containing chemotherapy in combination with a biologic agent

  * Inclusion Criteria for Cohort B:
* Disease progression during or following not more than two separate lines of treatment for mCRC that consisted of oxaliplatin, and irinotecan containing chemotherapy in combination with a biologic agent

Exclusion Criteria:

* Previous anticancer treatment within 4 weeks prior to initiation of study treatment
* Prior allogeneic stem cell or solid organ transplant
* Treatment with systemic immunostimulatory agents within 4 weeks prior to initiation of study treatment
* Use of any live vaccines against infectious diseases within 28 days of first dose.
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases
* Current treatment with anti-viral therapy for HBV
* Structurally unstable bone lesions suggesting impending fracture
* History or leptomeningeal disease
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan
* History of malignancy other than colorectal cancer within 2 years prior to screening, except for malignancies such as non-melanoma skin carcinoma or ductal carcinoma in situ
* Active tuberculosis
* Treatment with therapeutic oral or intravenous (IV) antibiotics within 2 weeks prior to initiating study treatment
* Severe infection within 4 weeks (28 days) prior to initiation of study treatment
* Significant cardiovascular disease, unstable or new onset of angina within 3 months prior to initiation of treatment, or myocardial infarction within 6 months prior to study treatment or unstable arrhythmia
* Major surgical procedures, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for major surgical procedure during the study
* Known allergy or hypersensitivity to any of the study drugs or their excipients
* Inability to swallow medications
* Malabsorption condition that would alter the absorption of orally administered medications
* Evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
* Prior treatment with an agent targeting the adenosine pathway
* Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain Barré syndrome, or multiple sclerosis

  * Exclusion Criteria for Cohorts A and B:
* Prior treatment with immune checkpoint blockade therapies including anti-cytotoxic T lymphocyte-associated protein-4, anti PD-1, and anti-PD-L1 therapeutic antibodies
* Mutation in the BRAF oncogene. Patients with unknown BRAF status will be required to undergo testing at a local laboratory and provide results at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2025-09-05 (Actual); Study Completion 2025-09-05 (Actual)

PRIMARY OUTCOMES:
Cohort A and B - Progression-free Survival (PFS) | From randomization until death from any cause (up to approximately 3-7 years)
  PFS according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, as assessed by the Investigator
Cohort C - Objective Response Rate (ORR) | From randomization until death from any cause (up to approximately 3-7 years)
  ORR according to RECIST v1.1, as assessed by the Investigator
Number of Participants With Treatment-emergent Adverse Events | Up to approximately 10 Months

SECONDARY OUTCOMES:
Cohorts A and B - Objective Response Rate (ORR) | From randomization until death from any cause (up to approximately 3-7 years)
  ORR according to RECIST v1.1 as assessed by the Investigator
Cohorts A, B, and C- Duration of Disease Response (DoR) | From randomization until death from any cause (up to approximately 3-7 years)
  DoR according to RECIST v1.1, as assessed by the Investigator
Cohorts A, B, and C- Disease Control Rate (DCR) | From randomization until death from any cause (up to approximately 3-7 years)
  DCR according to RECIST v1.1, as assessed by the Investigator
Cohorts A and B - Overall Survival (OS) | From randomization until death from any cause (up to approximately 3-7 years)
  OS according to RECIST v1.1, as assessed by the Investigator
Observed Maximum Concentration (Cmax) of Etrumadenant and its Metabolites | From randomization until death from any cause (up to approximately 10 months)
  Cycle 1 Day 1 and Cycle 2 Day 1
Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours [AUC(0-24)] of Etrumadenant and its Metabolites | Up to 24 hours following Day 1 Cycle 1 and Cycle 2 (each cycle is 28 days)
Trough Concentrations of Etrumadenant and its Metabolites | Multiple timepoints up to approximately 16 months
Cmax End of Infusion (EOI) of AB680 | At the end of infusion on Day 1 Cycle 1 and Cycle 2 (each cycle is 28 days)
Area Under the Plasma Concentration Versus Time Curve From Time Zero to 336 Hours [AUC(0-336)] of AB680 | Up to 336 hours following Day 1 Cycle and Cycle 2 (each cycle is 28 days)]
Trough Concentrations of AB680 | Multiple timepoints up to approximately 16 months
Cmax EOI of Zimberelimab | Multiple timepoints up to approximately 16 months
AUV(0-336) of Zimberelimab | Cycle 1 Day 1 up to 336 hours
Trough Concentrations of Zimberelimab | Multiple timepoints up to approximately 16 months
Number of Participants With Anti-Drug Antibodies to the Biologic Component(s) of Combination Therapy | Up to approximately 10 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Arcus Biosciences
Locations (44):
- United States (17):
  - Arizona Clinical Research Center Inc, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UCLA Hematology Oncology, Santa Monica, California
  - Yale Cancer Center, New Haven, Connecticut
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Ochsner Medical Center (OMC), New Orleans, Louisiana
  - American Oncology Partners of Maryland PA, Bethesda, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Comprehensive Cancer Centers Of Nevada, Las Vegas, Nevada
  - NYU Langone Medical Center - NYU Medical Oncology Associates, New York, New York
  - New York-Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Prisma Health-Upstate, Greenville, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Wisconsin School of Medicine, Madison, Wisconsin
- France (6):
  - Institut Bergonie - Centre Regional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - Centre Georges Francois Leclerc, Dijon
  - Hopital Hotel Dieu, Nantes
  - Hopital Saint Antoine, Paris
  - Groupe Hospitalier Pitie-Salpetriere-Centre De Recherche et de Medecine de l'Obesite, Paris
  - CHU la Miletrie, Poitiers
- Italy (6):
  - IRCCS - Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis, Castellana Grotte
  - Azienda Ospedaliero Universitaria Careggi-S.O.D. Patologia Medica, Florence
  - Azienda Ospedaliera Niguarda Ca' Granda, Milan
  - Instituto Europeo di Oncologia, Milan
  - Istituto Clinico Humanitas IRCCS, Rozzano
  - Universita di Siena - Azienda Ospedaliera Universitaria Senese-Policlincio Santa Maria Alle Scotte, Siena
- South Korea (8):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Bundang Hospital, Seoul
  - Seoul National University Hospital (SNUH), Seoul
  - Severance Hospital | Yonsei University Health System, Seoul
  - Asan Medical Center | University of Ulsan College of Medicine, Seoul
  - Samsung Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyungpook National University Chilgok Hospital, Seoul
- Spain (5):
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Complejo Hospitalario de Orense, Ourense
  - Clinica Universidad Navarra-Sede Madrid, Pamplona
  - Corporacio Sanitaria Parc Tauli, Sabadell
- United Kingdom (2):
  - Belfast City Hospital, Belfast, Northern Ireland
  - Aberdeen Royal Infirmary, Aberdeen, Scotland

IPD SHARING:
Plan to Share IPD: Yes
Arcus will provide access to individual de-identified participant data and related study documents (e.g., protocol, Statistical Analysis Plan [SAP], Clinical Study Report [CSR]) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions.
  For more information, please visit our website.
Supporting Information: Study Protocol, SAP, CSR
URL: https://trials.arcusbio.com/our-transparency-policy

REFERENCES:
- See also: ARC-9 - Public website — https://trials.arcusbio.com/study/?id=ARC-9